CLINICAL TRIAL: NCT07261163
Title: Obinutuzumab, Zanubrutinib, and Lenalidomide as First-Line Therapy for Mantle Cell Lymphoma: A Prospective, Single-Arm, Open-Label, Multicenter Study
Brief Title: Obinutuzumab, Zanubrutinib, and Lenalidomide in First-line Treatment of Mantle Cell Lymphoma
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Institute of Hematology & Blood Diseases Hospital, China (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IIT2025103
Record Dates: First submitted 2025-11-21; First posted 2025-12-03 (Actual); Last update posted 2025-12-03 (Actual); Status verified 2025-07

CONDITIONS: Mantle Cell Lymphoma
MeSH Terms: conditions — Lymphoma, Mantle-Cell | interventions — zanubrutinib; obinutuzumab; Lenalidomide; Immunotherapy, Adoptive

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- ZGR (Experimental)
  Interventions: Drug: Zanubrutinib; Drug: Obinutuzumab; Drug: Lenalidomide; Other: CAR-T Cell Therapy

INTERVENTIONS:
Drug: Zanubrutinib — Zanubrutinib 160 mg orally twice daily (bid), continuously administered. Used during the induction phase as part of the ZGR regimen for 6 cycles, and continued as maintenance therapy for up to 2 years. For patients not achieving complete response, treatment may be extended beyond 2 years until disease progression or intolerance.
Drug: Obinutuzumab — Obinutuzumab 1000 mg administered intravenously. Dosing schedule: Days 1, 8, and 15 of Cycle 1; Day 1 of each subsequent cycle starting from Cycle 2. Each cycle is 28 days. Administered as part of the ZGR induction regimen for 6 cycles.
Drug: Lenalidomide — Lenalidomide 20 mg orally once daily on Days 1-21 of each 28-day cycle. Administered during the induction phase as part of the ZGR regimen for 6 cycles. For maintenance, the dose is reduced to 10 mg once daily on Days 1-21 of each 28-day cycle, for a duration of 1 year.
Other: CAR-T Cell Therapy — For high-risk patients, CAR-T cell therapy is permitted after completion of the induction phase. Initiation of CAR-T therapy is followed by a 2-month recovery period before starting maintenance therapy with zanubrutinib and lenalidomide.

SUMMARY:
This is a prospective, open-label, single-arm clinical trial evaluating a treatment strategy for previously untreated Mantle Cell Lymphoma (MCL). The study will enroll patients who have not received prior systemic therapy for MCL. All patients will receive the ZGR induction regimen. Risk-adapted maintenance therapy will be applied: non-high-risk patients will receive lenalidomide and zanubrutinib maintenance for 1 and 2 years, respectively; high-risk patients will undergo CAR-T cell therapy followed by the same maintenance regimen. The primary objective is to assess the feasibility and preliminary efficacy of this treatment approach in the first-line setting of MCL.

ELIGIBILITY:
Inclusion Criteria:

1. Age between 18 and 80 years inclusive, both genders are eligible.
2. Histologically or cytologically confirmed diagnosis of Mantle Cell Lymphoma (MCL), with at least one measurable lesion according to Lugano criteria.
3. No prior systemic therapy for MCL.
4. Eastern Cooperative Oncology Group (ECOG) performance status of 0 to 2.
5. Adequate organ function, defined as:

   1. Hematologic function (without red blood cell or platelet transfusion, growth factor support, or medication correction within 14 days prior to enrollment):Absolute neutrophil count (ANC) ≥ 1 × 10⁹/L;Platelet count (PLT) ≥ 75 × 10⁹/L;
   2. Biochemical tests must meet the following criteria::

      Total bilirubin ≤ 2.0 × upper limit of normal (ULN);Alanine aminotransferase (ALT) and aspartate aminotransferase (AST) ≤ 2.0 × ULN;Creatinine clearance ≥ 30 mL/min, calculated by the Cockcroft-Gault formula;
   3. Cardiac function:Left ventricular ejection fraction (LVEF) ≥ 50% by echocardiogram.
6. Female subjects of childbearing potential must have a negative serum pregnancy test within 7 days prior to initiation of study treatment, and must agree to use a highly effective method of contraception (e.g., intrauterine device, hormonal contraception, or condom use) during the study and for 6 months after the last dose of study drug. Male subjects whose partners are of childbearing potential must be surgically sterile or agree to use effective contraception during the study and for 6 months after the last dose of study drug.
7. Willing and able to provide written informed consent and comply with the study follow-up requirements.

Exclusion Criteria:

1. Known central nervous system (CNS) involvement, including brain or meningeal lymphoma.
2. Congestive heart failure with New York Heart Association (NYHA) Class III or IV cardiac dysfunction.
3. History of other primary malignancies within the past 3 years, except for non-melanoma skin cancer, localized prostate cancer considered cured, cervical in situ carcinoma, or squamous intraepithelial lesion detected by PAP smear.
4. Prior treatment with investigational drugs.
5. Active systemic viral, bacterial, or fungal infection requiring antimicrobial therapy within 2 weeks prior to first administration of study drug.
6. Use of immunosuppressive agents within 7 days prior to first administration of study drug, except for intranasal or inhaled corticosteroids, or systemic corticosteroids at physiologic doses (i.e., ≤ 20 mg/day prednisone or equivalent).
7. History of hypersensitivity, allergic reactions, or adverse drug reactions:Severe hypersensitivity reaction to monoclonal antibodies;Allergy or intolerance to infusions;History of severe allergy to study drugs or premedication agents.
8. Physical or laboratory findings:Congenital or acquired immunodeficiency, such as active hepatitis B (HBV DNA ≥ 500 IU/mL), hepatitis C (positive HCV antibody and HCV-RNA above lower limit of detection), or co-infection with both HBV and HCV; Pregnant or breastfeeding women; subjects of childbearing potential unwilling or unable to use effective contraception; Known history of positive human immunodeficiency virus (HIV) test or acquired immunodeficiency syndrome (AIDS).
9. Any condition that, in the investigator's judgment, may impair subject safety or ability to comply with the study protocol.
10. Other conditions deemed unsuitable for enrollment by the investigator.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 37 (Estimated)
Dates: Start 2025-12-20 (Estimated); Primary Completion 2027-07-31 (Estimated); Study Completion 2029-07-31 (Estimated)

PRIMARY OUTCOMES:
complete response rate (CR) | up to the end of 6 cycles of treatment (each cycle is 28 days)
  To assess the complete response rate (CR) at the end of Induction therapy [Time Frame: up to the end of induction treatment

SECONDARY OUTCOMES:
Overall Response Rate (ORR) | up to the end of 6 cycles of treatment (each cycle is 28 days)
  Response Rate (ORR) is defined as the proportion of subjects who achieve CR or PR after Induction treatment
Duration of Response (DoR) | [Time Frame: up to 5 years]
  The length of time between the achievement of criteria for response to treatment (first documented complete or partial response) and the first documented relapse or progression.
Progression-free survival (PFS) | [Time Frame: up to 5 years]
  The time from the enrollment of a subject to the occurrence of (in any way) progression of disease or Death for any reason. patients with indeterminate recurrence or Death at the last follow-up, defined as the date of the last Investigation
Overall survival | [Time Frame: up to 10 years]
  The time from subject enrollment to Death caused by any reason. for patients lost to follow-up, the time of the lastfollow-up; for patients still alive at the end of study, the date of the end of follow-up.
The safety | Time Frame: up to 5 years
  Incidence of adverse events, serious adverse events and significant adverse event

CONTACTS AND LOCATIONS:
Locations (1):
- Institute of Hematology & Blood Diseases Hospital, Tianjin, Tianjin Municipality, China

IPD SHARING:
Plan to Share IPD: No